CLINICAL TRIAL: NCT01800435
Title: Whole Blood Clot Stability and Thrombin Generating Capacity Following Treatment With Bypassing Agents (BPA) With and Without and Tranexamic Acid (TXA) in Haemophilia A Patients With inhibitor-an In-vivo Prospective Crossover Study
Brief Title: A Comparison Study of Bypassing Agent Therapy With and Without Tranexamic Acid in Haemophilia A Patients With Inhibitor
Acronym: BPATXAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Pål Andre Holme, MD PhD, Oslo University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EudraCTnr. 2010-022668-11; 2010-022668-11 (EudraCT Number)
Record Dates: First submitted 2013-02-15; First posted 2013-02-27 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Hereditary Factor VIII Deficiency Disease With Inhibitor
MeSH Terms: interventions — Tranexamic Acid; recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aPCC, aPCC + TXA (Active Comparator): aPCC 75IU/kg i.v aPCC 75IU/kg i.v +TXA 20mg/kg
  Interventions: Drug: aPCC, aPCC + TXA; Drug: rFVIIa, rFVIIa + TXA
- rFVIIa, rFVIIa + TXA (Active Comparator): rFVIIa 90 µg/kg i.v rFVIIa 90 µg/kg i.v + TXA 20 mg/kg
  Interventions: Drug: aPCC, aPCC + TXA; Drug: rFVIIa, rFVIIa + TXA

INTERVENTIONS:
Drug: aPCC, aPCC + TXA — Feiba 75 IU/kg i.v Feiba 75 IU/kg i.v +Cyklokapron 20 mg/kg p.o
  Other Names: Feiba i.v; Feiba i.v + Cyklokapron
Drug: rFVIIa, rFVIIa + TXA — NovoSeven 90 µg/kg i.v NovoSeven 90 µg/kg i.v + Cyklokapron 20 mg/kg
  Other Names: NovoSeven 90 µg/kg i.v; NovoSeven 90 µg/kg i.v + Cyklokapron 20 mg/kg

SUMMARY:
Activated prothrombin complex concentrate (aPCC) and recombinant activated factor VII (rFVIIa) are the only two drugs that are available to treat bleeds in haemophilia A patients with high titer inhibitors. However, management of bleeds in these patients can be challenging due to variation in response and lack of standardized methods to monitor the effect. We hypothesized that significant increase in whole blood clot stability could be achieved when tranexamic acid was given concomitantly with bypassing-agents while thrombin generation remains unaffected. In this prospective crossover study the effect of aPCC and rFVIIa with and without TXA on clot stability and thrombin generation capacity (ETP) were studied, using thromboelastography (ROTEM) and thrombin generation assay (TGA), respectively. In addition, the risk of thrombosis and disseminated intravascular coagulation (DIC) was assessed.

DETAILED DESCRIPTION:
Patients receive the first day aPCC (75IU/kg) and aPCC in addition to TXA (20mg/kg orally) the second day. After a 14 days washout period they crosse over using rFVIIa (90 µg/kg) otherwise the same experimental setup. Blood sampling is performed at baseline, 15, 30, 60, 120, 180 and 240 minutes post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia patients with high titer inhibitors or high-responding inhibitors, aged between 18-65 and no history of aspirin or NSAID use within the last 14 days were eligible for the study.

Exclusion Criteria:

* Patients with renal failure, liver disease, infected with immune deficiency virus (HIV), platelet count <150x109/L, acquired haemophilia, ongoing bleeding, hypersensitivity to TXA or a history of arterial or venous thrombosis were excluded from the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Clot stability and thrombin generation capacity following treatment with bypassing agents with and without tranexamic acid. | 2 years
  MCF (maximum clot formation/mm x 100-1), AUC (area under the elasticity curve AUC, mm• 100 s-1) were used as the primary outcome measures for evaluating clot stability and (ETP) the coagulable state.

SECONDARY OUTCOMES:
DIC or thrombosis events associated with different treatment regimens. | 2 years
  DIC parameters such as aPTT, PT/INR, platelet count, fibrinogen and D-dimer with the scoring system proposed by the International Society of Thrombosis and Haemostasis were used to monitor DIC in addition to common clinical signs associated with DIC were records. Symptoms or clinical signs of thrombosis such as dyspnea, chest pain, legg swelling or discomfort/pain were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: PÅL A Holme, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway